CLINICAL TRIAL: NCT03547375
Title: Clinical Study of Apatinib in the Treatment of Advanced Ovarian Cancer After the Failure of Standard Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHTH-102
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment group (Experimental): Apatinib 500mg/d po,28 days as one cycle
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg/d po,28 days as one cycle

SUMMARY:
To Observe and Evaluate the Efficacy and Safety of Apatinib in Patients With Advanced Ovarian Cancer After the Failure of Standard Chemotherapy

DETAILED DESCRIPTION:
Eligible patients will receive apatinib 500mg/d po until disease progression or intolerable toxicity or patients withdrawal of consent after the failure of chemotherapy or radiotherapy

ELIGIBILITY:
Inclusion Criteria:

1. ovarian cancer confirmed by pathology;
2. At least one measuring lesion (RECIST 1.1) or ascites (B ultrasound);
3. Patients with advanced ovarian cancer who failed in standard treatment. Note: Advanced ovarian cancer with recurrence of platinum-resistant drug and having no possibility of surgery
4. Baseline blood routine and biochemical indicators meet the following criteria:

   ① ANC ≥ 1.5 × 109 / L;
   * HB ≥ 90g / L;

     * PLT ≥ 100 × 109 / L; ④ ALB≥30g / L;

       * TBIL≤1.5 times the upper limit of normal (ULN); ⑥ ALT and AST<2 × ULN; ⑦ Plasma Cr<1.5 × ULN
5. No blood transfusion , blood products, G-CSF and other hematopoietic stimulation factors were used in 14 days ;
6. The expected survival time is longer than 3 months;
7. The pregnancy test (serum or urine)should be carried out for women in childbearing age before 7 days into the group and the results were negative, and willing to use appropriate methods of contraception during the test and after 8 weeks out of group
8. The subjects volunteered to participate in this study, signed informed consent, followed up with good compliance .

Exclusion Criteria:

1. Allergies to apatinib and/or its excipients
2. People with high blood pressure and antihypertensive drug treatment can not drop to normal range (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), with level-1 above coronary heart disease, arrhythmia over class I (including QTc lengthened men > 450 ms, women > 470 ms).
3. According to NYHA standard, Ⅲ - Ⅳ cardiac insufficiency, or LVEF < 50%;
4. Various factors that affect oral drugs (such as inability to swallow, nausea, vomiting, chronic diarrhea, intestinal obstruction, etc.);
5. Patients with a clear tendency of gastrointestinal bleeding, including the following situations: local active ulcer lesions, and fecal occult blood (++); Patients with black stool and hematemesis in 2 months;
6. Abnormal coagulation function (INR>1.5, APTT>1.5 ULN), with bleeding tendency;Hereditary or acquired bleeding and thrombosis tendencies (such as hemophilia,coagulation dysfunction, thrombocytopenia, hypersplenism, etc.);
7. Long-term unhealed wounds or fractures; Major surgery or severe traumatic injury, fracture or ulcer in 4 weeks;
8. With abdominal fistula, gastrointestinal perforation or abdominal abscess;Active patients with HBV or HCV;
9. Active brain metastases, meningitis, cancer patients with spinal cord compression, CT or MRI examination revealed brain or soft meningeal disease (21 days before the drug treatment; the symptoms of patients with stable brain metastases can into the group, but need to be confirmed by the cerebral MRI, CT or vein imaging evaluation no cerebral hemorrhage).
10. CT or MRI showed that the tumor lesion was less than 5 mm away from the large vessel, or the lesion invaded local large vessels;
11. Pregnant or lactating women;
12. Patients with a history of psychotropic substance abuse or have mental disorders;
13. According to the researchers' judgment, patients who have serious harm to the patient's safety or affect the patients for completing the research;
14. Subjects considered inappropriate by the researchers.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | An expected average of 12 weeks
  The time from the beginning of treatment to observing the progression of the disease or the death of any cause